CLINICAL TRIAL: NCT01943695
Title: Optimal Timing Trial: Randomized Trial of Supervised Aerobic Training During or After Chemotherapy for Operable Breast Cancer
Brief Title: Supervised Aerobic Training During or After Chemotherapy for Operable Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-178
Record Dates: First submitted 2013-07-31; First posted 2013-09-17 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Exercise; Chemotherapy; 15-178
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aerobic Training During Chemotherapy (Experimental): The ultimate goal is for participants to complete approximately 3 exercise sessions week of non-linear aerobic training an intensity of at 55% to 100% of the individually determined exercise capacity VO2peak), concurrent with chemotherapy. VO2peak will be determined by the CPET performed at baseline. The weekly exercise will be achieved via 3 individual aerobic training sessions ranging from approximately 20-45 min/session. All sessions are required to be supervised unless otherwise specified by EP discretion.
  Interventions: Behavioral: Aerobic Training
- Aerobic Training After Chemotherapy (Experimental): The ultimate goal is for participants to complete approximately 3 exercise sessions week of non-linear aerobic training at an intensity 55% to 100% of the individually determined exercise capacity (VO2peak), after the completion of chemotherapy. VO2peak will be determined by the CPET performed at midpoint, or pre-surgery for neoadjuvant patients. For patients receiving adjuvant therapy, (except those who have additional surgery after chemotherapy), the aerobic training intervention must begin within 2 weeks of the patient's midpoint CPET. For patients receiving neoadjuvant or adjuvant therapy and have additional surgery after chemotherapy, the aerobic training intervention will begin within approximately 6 weeks of surgery, per the discretion of the treating physician. The weekly exercise will be achieved via 3 individual aerobic training sessions ranging from approximately 20-45 min/session. All sessions are required to be supervised unless otherwise specified by EP discretion.
  Interventions: Behavioral: Aerobic Training
- Continuous Aerobic Training (Experimental): The ultimate goal is for participants to complete 3 exercise sessions week of non-linear aerobic training at 55% to 100% of the individually determined exercise capacity (VO2peak), during and after chemotherapy. For patients receiving adjuvant therapy (except those who have additional surgery after chemotherapy), VO2peak will be determined by the CPETs performed at baseline and midpoint. For patients receiving neoadjuvant or adjuvant therapy and have additional surgery after chemotherapy, VO2peak will be determined by the CPETs or at baseline, pre- surgery, and post-surgery. The weekly exercise will be achieved via 3 individual aerobic training sessions ranging from approximately 20-45 min/session. All sessions are required to be supervised unless otherwise specified by EP discretion.
  Interventions: Behavioral: Aerobic Training
- General Physical Activity Group (Experimental): Patients will receive a home-based, general physical activity program. Specifically, all patients assigned to general physical activity will receive an initial, consultation with a staff exercise physiologist outlining a structured home-based aerobic walking program with a goal up to 150 minutes per week outside of their normal daily activity. Patients can be provided with a fitness tracker (e.g. FitBit) to evaluate exercise duration and intensity. Patients may also be provided with an exercise log to record type, duration, and average heart rate during sessions. The exercise log is provided as a guidance tool and may be, although is not required to be, returned to study staff. Staff exercise physiologists will contact patients to check progress, and answer questions.
  Interventions: Behavioral: Educational Information; Behavioral: Supervised Home Based Training

INTERVENTIONS:
Behavioral: Aerobic Training
  Other Names: exercise, breast cancer, therapy.
  Arms: Aerobic Training After Chemotherapy; Aerobic Training During Chemotherapy; Continuous Aerobic Training
Behavioral: Educational Information — Subjects will be given material regarding cancer and it's impact.
  Arms: General Physical Activity Group
Behavioral: Supervised Home Based Training — Patients that elect supervised home based training platform or plan to complete unsupervised training sessions will receive a study kit which includes a heart rate monitor, blood pressure cuff, treadmill and tablet to complete aerobic training requirements. The study kit will be given to the patient upon completion of their baseline testing. The treadmill will be shipped to the patient's home and coordinated by the Ex Onc group. The treadmills are MSK owned equipment that will be deployed to the patient's homes via the vendor TechnoGym. A member of Ex Onc will provide an orientation session for the patient to set up all study kit items. If there is a delay in the patient receiving the treadmill , or any other unforeseen circumstance, patients may be assigned a temporary unsupervised training program until the treadmill is delivered.
  Arms: General Physical Activity Group

SUMMARY:
The purpose of this study is to compare the effects of aerobic exercise training during and after chemotherapy for women who have recently been diagnosed with early-stage breast cancer.

The participant will be instructed to self-report the session information to ExOnc staff at or before their next scheduled visit. If the participant's next scheduled visit is greater than 72 hours following an unsupervised session, ExOnc staff may reach out to the participant to retrieve the session information. Unsupervised session details will be source documented by ExOnc staff.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-80 years
* Female
* MSK histologically confirmed early-stage operable breast cancer
* Scheduled to receive chemotherapy in the neoadjuvant or adjuvant setting
* ECOG status of 0 or 1
* Performing less than 150 minutes of structured moderate-intensity or strenuous intensity exercise per week
* If a female of child-bearing potential, must not be pregnant or planning to become pregnant during the study.

  a. Women < 50 years old must have a negative pregnancy test (urine HCG or serum βHCG) within 2 weeks of beginning chemotherapy.
* Able to complete an acceptable baseline cardiopulmonary exercise test (CPET), in the absence of high risk ECG findings or other inappropriate response to exercise as determined by the investigator.
* Able to achieve an acceptable peak baseline CPET, as defined by any of the following criteria:

  * Achieving a plateau in oxygen consumption, concurrent with an increase in power output;
  * A respiratory exchange ratio ≥ 1.10;
  * Attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted HRmax [HRmax = 220-Age[years]);
  * Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.
* Willingness to be randomized to one of the study arms

Exclusion Criteria:

* Presence of any other concurrent, actively treated malignancy
* History of any other malignancy treated within the past 3 years (other than non-melanoma skin cancer)
* Presence of metastatic disease
* Any of the following contraindications to cardiopulmonary exercise testing:
* Acute myocardial infarction within 3-5 days of any planned study procedures)
* Unstable angina
* Uncontrolled arrhythmia causing symptoms or hemodynamic compromise;
* Recurrent syncope
* Active endocarditis
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures;
* Thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Respiratory failure
* Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis) or
* Room air desaturation at rest ≤ 85%
* Mental impairment leading to inability to cooperate.
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the participant a poor candidate for the trial

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-01; Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in VO2 peak (functional capacity) | during chemotherapy 3-6 months depending on treatment recommendations
  To determine the optimal timing of aerobic activity, relative to an attention-control group, on exercise capacity in a breast cancer setting. This will be evaluated using an electronic motorized treadmill test with 12-lead ECG monitoring (Mac® 5000, GE Healthcare) performed by certified exercise physiologists.

SECONDARY OUTCOMES:
Quality of Life measured by questionnaire during and after Chemotherapy | at baseline, mid-point (12 weeks approximately) , and follow-up (24 weeks approximately) testing
  Determine the effects on patient-reported outcomes. Time frame can vary based on individual length of chemotherapy.
Sleeping patterns as measured by questionnaire during and after Chemotherapy | at baseline, mid-point (12 weeks approximately) , and follow-up (24 weeks approximately) testing
  Determine the effects on patient-reported outcomes. Time frame can vary based on individual length of chemotherapy.
Depression scale during and after Chemotherapy | at baseline, mid-point (12 weeks approximately) , and follow-up (24 weeks approximately) testing
  Determine the effects on patient-reported outcomes. Time frame can vary based on individual length of chemotherapy.
Physical activity recall during and after Chemotherapy | at baseline, mid-point (12 weeks approximately) , and follow-up (24 weeks approximately) testing
  Determine the effects on patient-reported outcomes. Time frame can vary based on individual length of chemotherapy.
Skeletal Muscle Function | at baseline, mid-point (12 weeks approximately) , and follow-up (24 weeks approximately) testing
  To examine the physiological mediators of the exercise training - exercise capacity relationship (e.g., skeletal muscle function as assessed by a muscle biopsy)performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Iyengar NM, Scott JM, Lee J, Lavery JA, Foug KL, Lee CP, Michalski MG, Chun SS, Harrison J, Moskowitz CS, Jones LW. Effects of exercise therapy on chemotherapy delivery and response in primary breast cancer: A secondary analysis of a randomized trial. Cancer. 2025 Jan 1;131(1):e35575. doi: 10.1002/cncr.35575. Epub 2024 Sep 22. PMID 39306704
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/